CLINICAL TRIAL: NCT00462644
Title: A Single Dose of Etomidate During Rapid Sequence Induction in Trauma Patients Causes Significant Adrenocortical Insufficiency: A Prospective Randomized Study
Brief Title: Evaluation of Etomidate on Adrenal Function in Trauma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Responsible Party: Vicente A. Mejia, MD, University of Tennessee College of Medicine, Chattanooga
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 05-050
Record Dates: First submitted 2007-04-17; First posted 2007-04-19 (Estimated); Results first posted 2009-11-11 (Estimated); Last update posted 2010-02-23 (Estimated); Status verified 2010-02

CONDITIONS: Adrenal Insufficiency
Keywords: adrenal insufficiency; etomidate; rapid sequence induction
MeSH Terms: conditions — Adrenal Insufficiency | interventions — Etomidate; Succinylcholine; Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Etomidate (Active Comparator): Etomidate Group patients were randomized to receive etomidate 0.3mg/kg IV plus succinylcholine 1mg/kg IV for RSI medications
  Interventions: Drug: RSI sedation with etomidate/succinylcholine
- Fentanyl-Midazolam (Active Comparator): Fentanyl-Midazolam Group patients were randomized to receive 100ug fentanyl IV, plus 5 mg midazolam IV, plus 1mg/kg succinylcholine IV for RSI medications.
  Interventions: Drug: RSI sedation with fentanyl/midazolam/succinylcholine

INTERVENTIONS:
Drug: RSI sedation with etomidate/succinylcholine — etomidate 0.3 mg/kg IV plus succinylcholine 1 mg/kg IV
  Arms: Etomidate
Drug: RSI sedation with fentanyl/midazolam/succinylcholine — 100 micrograms fentanyl IV, plus 5 mg midazolam IV, plus 1 mg/kg succinylcholine IV
  Arms: Fentanyl-Midazolam

SUMMARY:
Trauma patients are at increased risk for adrenal function insufficiency. A commonly used agent for rapid sequence intubation (RSI) is known to decrease adrenal function. We want to determine the incidence of adrenocortical insufficiency and its significance during the first 24 hours of resuscitation following RSI in trauma patients.

DETAILED DESCRIPTION:
The study will have two arms. Patients on one arm will be assigned to receive etomidate (0.3 mg/kg) and succinylcholine (1mg/kg) for RSI. Patients on the other arm will receive standard therapy at this institution which consists of Versed (generic name midazolam) (5 mg) plus fentanyl (100 mcgs) as well as succinylcholine for RSI. Both drug regimens have a rapid onset, short duration and short half-life.

Patients will be randomly assigned to one arm of the study. The trauma nurse emergency room responders, intensive care unit staff, or helicopter crew will pull a study envelope which will contain a randomization to either the etomidate arm or standard therapy arm. The numbers will correspond to a log, delineating which medication is given. The nurse will document the medication as RSI Study Drug - etomidate or RSI Study Drug - standard and the randomization packet number (ie, RSI Study Drug, etomidate, #1, RSI Study Drug, standard, #2, etc.) and will document the patient's name and medical record number on the study log in either the helicopter or the ER Resuscitation Bay.

Baseline cortisol level will be drawn prior to RSI. An additional cortisol level will be drawn 4-6 hours later. Following this level, a cortrosyn stimulation test will be performed by giving 0.25 mg cortrosyn IV and rechecking a cortisol level in 60 minutes. Adrenal insufficiency will be defined as a baseline cortisol level of <15 or an increase in cortisol of <9 after cortrosyn administration. Patients will be monitored for 24 hours for hemodynamics, IV fluid administration , and use of vasopressors. Patient will be resuscitated to adequate mean arterial blood pressure and urine output. Any patient found to be adrenal insufficient will be treated with hydrocortisone 50 mg IV every 6 hours.

ELIGIBILITY:
Inclusion Criteria:

* Trauma mechanism of injury
* Patient requires rapid sequence induction for ventilatory support

Exclusion Criteria:

* <18 years old
* Prisoners
* Pregnant women
* Patients with a history of adrenal insufficiency
* Patients with adrenal trauma documented by CT scan
* Patients receiving corticosteroids in the previous year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-02; Primary Completion 2006-08 (Actual); Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vicente A Mejia, MD, Principal Investigator — University of Tennessee
Locations (1):
- Erlanger Medical Center, Chattanooga, Tennessee, United States

REFERENCES:
- [Result] Hildreth AN, Mejia VA, Maxwell RA, Smith PW, Dart BW, Barker DE. Adrenal suppression following a single dose of etomidate for rapid sequence induction: a prospective randomized study. J Trauma. 2008 Sep;65(3):573-9. doi: 10.1097/TA.0b013e31818255e8. PMID 18784570

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult trauma patients admitted to Erlanger Health System's Level I trauma center requiring rapid sequence induction were randomized to one of two approved drug treatment regimens.
Pre-assignment Details: 72 hour waiver of consent granted by the Institutional Review Board (IRB)
Period: Overall Study
Arm/Group | Etomidate | Fentanyl-Midazolam
Started | 18 | 12
Completed | 18 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Etomidate | Fentanyl-Midazolam | Total
Number analyzed (Participants) | 18 | 12 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0.0
  Between 18 and 65 years | 14 | 10 | 24.0
  >=65 years | 4 | 2 | 6.0
Age Continuous [Mean (Standard Deviation); unit: years] | 41.8 (24.5) | 43.9 (19.5) | 42.6 (22.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 3 | 11.0
  Male | 10 | 9 | 19.0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 12 | 30.0

OUTCOME MEASURES:

1. Primary Outcome: Cortisol Levels Pre and Post Rapid Sequence Induction and Cortisol Stimulation Test
Time Frame: pre RSI, 4-6 hours post RSI, and again 60 mins later following ACTH stimulation test
Reporting Status: Not Posted

2. Secondary Outcome: Hospital Length of Stay
Description: days from admission to hospital discharge
Time Frame: time to hospital discharge in days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Etomidate | Fentanyl-Midazolam
Number analyzed (Participants) | 18 | 12
days | 13.9 (9.5) | 6.4 (4.4)
Statistical Analysis 1: Comparison: Etomidate vs Fentanyl-Midazolam; Test type: Superiority or Other; p = 0.007, t-test, 2 sided

3. Secondary Outcome: Intensive Care Unit (ICU) Length of Stay
Description: ICU length of stay in days
Time Frame: time from hospital admission to transfer out of ICU to floor bed
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Etomidate | Fentanyl-Midazolam
Number analyzed (Participants) | 18 | 12
days | 8.1 (7.2) | 3.0 (2.4)
Statistical Analysis 1: Comparison: Etomidate vs Fentanyl-Midazolam; Test type: Superiority or Other; p = 0.011, t-test, 2 sided

4. Secondary Outcome: Ventilator Days
Time Frame: time from intubation to extubation
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Etomidate | Fentanyl-Midazolam
Number analyzed (Participants) | 18 | 12
days | 6.3 (6.5) | 1.5 (0.8)
Statistical Analysis 1: Comparison: Etomidate vs Fentanyl-Midazolam; Test type: Superiority or Other; p = 0.007, t-test, 2 sided

5. Primary Outcome: Postintubation Cortisol (Baseline Cortisol Level)
Description: cortisol level after randomization and rapid sequence induction
Time Frame: postintubation (baseline cortisol level)
Measure: Mean (Standard Deviation); unit: micrograms/dL
Arm/Group | Etomidate | Fentanyl-Midazolam
Number analyzed (Participants) | 18 | 12
micrograms/dL | 18.2 (8.4) | 27.9 (13.4)
Statistical Analysis 1: Comparison: Etomidate vs Fentanyl-Midazolam; Normality was tested using the Kolmogorow-Smirnov test; Test type: Superiority or Other; p = 0.022, t-test, 2 sided

6. Primary Outcome: Change in Baseline Cortisol
Description: change from baseline cortisol (drawn prior to RSI) to 2nd cortisol level (4-6hrs after RSI, but before stim test)
Time Frame: 4-6hr after RSI
Measure: Mean (Standard Deviation); unit: micrograms/dL
Arm/Group | Etomidate | Fentanyl-Midazolam
Number analyzed (Participants) | 18 | 12
micrograms/dL | -12.8 (9.6) | 1.1 (7.6)
Statistical Analysis 1: Comparison: Etomidate vs Fentanyl-Midazolam; Test type: Superiority or Other; p = 0.003, t-test, 2 sided

7. Primary Outcome: Cortisol Level 60 Minutes After Cortisol Stimulating Test (CST)
Time Frame: 60 minutes after administration of cotrosyn
Measure: Mean (Standard Deviation); unit: micrograms/dL
Arm/Group | Etomidate | Fentanyl-Midazolam
Number analyzed (Participants) | 18 | 12
micrograms/dL | 22.91 (10.4) | 39.09 (10.8)
Statistical Analysis 1: Comparison: Etomidate vs Fentanyl-Midazolam; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

8. Secondary Outcome: Number of Deaths
Description: deaths
Time Frame: death in hospital
Measure: Number; unit: participants
Arm/Group | Etomidate | Fentanyl-Midazolam
Number analyzed (Participants) | 18 | 12
participants | 2 | 0

ADVERSE EVENTS:
Time Frame: from intubation until hospital discharge
Description: Two deaths occurred during hospitalization, but were not due to any study procedures. Deaths were due to trauma injuries sustained in conjunction with pre-existing conditions.
Arm/Group | Etomidate | Fentanyl-Midazolam
Serious Adverse Events (participants affected / at risk) | 2/18 | 0/12
Other Adverse Events (participants affected / at risk) | 0/18 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etomidate (N=18) | Fentanyl-Midazolam (N=12)
death (Cardiac disorders) | 2 (2) | 0 (0) — deaths occurred during hospitalization, but were not due to any study procedures.

LIMITATIONS AND CAVEATS:
Small trial most likely underpowered; large number of exclusions; other limitations discussed in published paper (PMID: 18784570).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No